CLINICAL TRIAL: NCT04997928
Title: Predicting The Prognosis Of Covid-19 Patients With Circulating Inflammatory and Coagulation Markers
Brief Title: PAI-1 Levels and Predicting Covid-19 Patients' Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nazlı ERCAN, Specialist Doctor, Saglik Bilimleri Universitesi
Other Study IDs: COVID19PAI-1
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Covid-19 Positivity Confirmed With PCR Positivity in the Nasopharyngeal Swab; Symptomatic Covid -19 Positive Patients Who Require Hospitalization; Patients Who Did Not Vaccinate Against Covid-19; Patients Among 20 to 90 Years of Age; Healthy Control Patients of the Same Age
Keywords: Covid-19; Polymerase Chain Reaction; Plasminogen activator inhibitor 1; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — After all four groups of patients have given their consent for the study, a sample of 5cc blood will be obtained once for the PAI-1 analysis. The sample will be centrifuged for around 5 minutes at 3000 rpm before being frozen at -70 degrees. The blood sample will be dissolved under proper conditions after a sufficient number of participants has been reached. The researchers will provide the ELISA kits for the study, and laboratory services will be purchased from outside the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (n=20; with mild symptoms): Group 1 (n=20; with mild symptoms)
  * Covid positive patients with mild symptoms who required to be hospitalized,
  * Symptomatic (fever, cough, weakness, joint pain, etc.) new patients who apply to the Covid clinic for the first time,
  * Patients with stable vital signs and/or SpO2 ≥92% in room air, no radiological signs of lung involvement or mild pneumonia,
  * Patients who have not been started on steroid therapy and who have not yet received anticoagulant therapy.
  Interventions: Other: Serum PAI-1 alpha analysis.
- Group 2 (n=20; with moderate symptoms): Group 2 (n=20; with moderate symptoms)
  * Patients who are positive for Covid 19 and admitted to the covid clinic for the first time;
  * Radiologically moderate pneumonia findings and/or SpO2=88-92% in room air,
  * Patients who have not been started antiviral, steroid, and anticoagulant treatment.
  Interventions: Other: Serum PAI-1 alpha analysis.
- Group 3 (n=20; with severe symptoms): Group 3 (n=20; with severe symptoms)
  * Patients who are currently hospitalized in the Covid clinic,
  * Patients with radiological findings of severe pneumonia or ARDS and/or high FiO2 requirement due to respiratory failure.
  * Patients of this group may have received antiviral, anticoagulant, and/or steroid and/or biologic agent treatment.
  Interventions: Other: Serum PAI-1 alpha analysis.
- Group 4 (n=20; Control group): Group 4 (n=20; Control group)
  * The control group will be composed of healthy adult individuals applying to adult allergy outpatient clinics on a voluntary basis.
  * Patients who have not been previously diagnosed with Covid-19 and have not vaccinated against Covid-19,
  * The control patients will be matched with the study groups according to age, gender, and BMI.
  Interventions: Other: Serum PAI-1 alpha analysis.

INTERVENTIONS:
Other: Serum PAI-1 alpha analysis. — After all four groups of patients have given their consent for the study, a sample of 5cc blood will be obtained once for the PAI-1 analysis.

SUMMARY:
The primary aim of our study is to understand the effects of Covid-19 disease on vascular inflammation and coagulation cascade, and secondarily, to investigate its utility in predicting disease prognosis by analyzing serum PAI-1 levels in patients with different severity. The study is planned as a prospective, cross-sectional study that will include patients admitted to Covid-19 services between January 18, 2021, and August 30, 2021. A total of 80 volunteers will be enrolled in the trial whose age, gender, and BMI are planned to be matched.The study will be conducted on four groups. Group 1 (n=20; with mild symptoms), Group 2 (n=20; with moderate symptoms), Group 3 (n=20; with severe symptoms) and Group 4 (n=20; Control group).

All participants who accepted the study will have their sociodemographic data, medical history, and vital signs (respiratory rate, saturation, temperature, and blood pressure values) recorded at the start of the study. The pulmonologist in the study will also classify the patient group's chest X-ray and chest tomography findings and the thymus gland dimensions. After all four groups of patients have given their consent for the study, a sample of 5cc blood will be obtained once for the PAI-1 analysis.

DETAILED DESCRIPTION:
The study is planned as a prospective, cross-sectional study that will include patients admitted to Covid-19 services between January 18, 2021, and August 30, 2021. A total of 80 volunteers will be enrolled in the trial whose age, gender, and BMI are planned to be matched. The study will be conducted on four groups.

Group 1 (n=20; with mild symptoms)

* Covid positive patients with mild symptoms who required to be hospitalized,
* Symptomatic (fever, cough, weakness, joint pain, etc.) new patients who apply to the Covid clinic for the first time,
* Patients with stable vital signs and/or SpO2 ≥92% in room air, no radiological signs of lung involvement or mild pneumonia,
* Patients who have not been started on steroid therapy and who have not yet received anticoagulant therapy.

Group 2 (n=20; with moderate symptoms)

* Patients who are positive for Covid 19 and admitted to the covid clinic for the first time;
* Radiologically moderate pneumonia findings and/or SpO2=88-92% in room air,
* Patients who have not been started antiviral, steroid, and anticoagulant treatment.

Group 3 (n=20; with severe symptoms)

* Patients who are currently hospitalized in the Covid clinic,
* Patients with radiological findings of severe pneumonia or ARDS and/or high FiO2 requirement due to respiratory failure.
* Patients of this group may have received antiviral, anticoagulant, and/or steroid and/or biologic agent treatment.

Group 4 (n=20; Control group)

* The control group will be composed of healthy adult individuals applying to adult allergy outpatient clinics on a voluntary basis.
* Patients who have not been previously diagnosed with Covid-19 and have not vaccinated against Covid-19,
* The control patients will be matched with the study groups according to age, gender, and BMI.

All participants who accepted the study will have their sociodemographic data, medical history, and vital signs (respiratory rate, saturation, temperature, and blood pressure values) recorded at the start of the study. The pulmonologist in the study will also classify the patient group's chest X-ray and chest tomography findings, as well as the thymus gland dimensions. After all four groups of patients have given their consent for the study, a sample of 5cc blood will be obtained once for the PAI-1analysis. The sample will be centrifuged for around 5 minutes at 3000 rpm before being frozen at -70 degrees. The blood sample will be dissolved under proper conditions after a sufficient number of participants has been reached. The researchers will provide the ELISA kits for the study, and laboratory services will be purchased from outside the hospital. Due to Covid-19 disease, white blood cell, neutrophil, lymphocyte, and platelet counts, liver enzymes (AST, ALT, LDH), sodium, total protein, albumin, aPTT, PTZ, INR, D-Dimer, and fibrinogen levels will be recorded in the patient case report form, as well as CRP, IL-6, and ferritin levels, which are routinely requested from patients during their hospitalization. No treatment other than the treatments specified in the Covid-19 guidelines of the Ministry of Health will never be applied to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 20 years of age and older, having Covid-19 PCR positivity in the nasopharyngeal swab and showing symptoms of Covid-19 (fever, cough, dyspnea, joint pain, etc.) with or without involvement in lung imaging.
2. Patients may have hypertension disease and type II diabetes mellitus (occurring less than 5 years, diet and/or insulin-regulated).
3. HbA1C levels of all participants (HbA1C < 6.4%) will be studied to confirm if any patient in the study or control groups has unregulated DM or undiagnosed overlooked DM. Diabetic patients with an HbA1C level above 6.4% will be excluded from the study.
4. Enrolled patients have to have a diagnostic chest X-ray and/or HRCT. (Participants will be subjected to radiological classification and scoring according to lung involvement such as ground-glass opacity.)

Exclusion Criteria:

* Patients who are considered to have previous vascular endothelial damage due to secondary causes such as history of thrombosis, thrombophlebitis and/or thromboembolism,
* Presence of active cancer, history of chemotherapy, radiotherapy or bone marrow transplantation,
* Presence or history of autoimmune, connective tissue diseases, vasculitis (autoimmune thyroiditis, Crohn's, ulcerative colitis, SLE, Sjogren's disease, etc.),
* Familial inherited hereditary diseases (Hemophilia, Mediterranean anemia, FMF, Thalassemia major etc.)
* Patients with chronic renal failure and/or requiring dialysis,
* Presence of acquired/congenital immunodeficiency,
* Patients who are receiving immunosuppressive or biologic drug therapy,
* Patients receiving treatment with a diagnosis of bronchial asthma,
* Type 1 or type 2 diabetes mellitus patients with HbA1C levels > 6.4%
* Patients with diabetes for more than 5 years or currently taking oral insulin-sensitizing drugs (biguanides; metformin)
* Patients using antithrombotic (Clopidogrel, low-dose aspirin, etc.) and anticoagulant (LMWH, Warfarin, etc.) agents due to comorbid disease at the time of diagnosis.
* Patients using ACE inhibitors such as lisinopril as an antihypertensive agent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: patients who are 20 years of age and older, having Covid-19 PCR positivity in the nasopharyngeal swab and showing symptoms of Covid-19 (fever, cough, dyspnea, joint pain, etc.) with or without involvement in lung imaging. A total of 80 volunteers will be enrolled in the trial whose age, gender, and BMI are planned to be matched.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum PAI-1 levels of Covid-19 patients | Blood sample collection is limited to up to 32 weeks and laboratory studies will be completed up to one week.
  To understand the effects of Covid-19 disease on vascular inflammation and coagulation cascade.

SECONDARY OUTCOMES:
Serum PAI-1 levels of Covid-19 patients | Up to 32 weeks for blood sample collection and up to one week for laboratory analysis.
  To investigate PAI-1 utility in predicting disease prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgür Kartal, MD, Study Chair — University of Health Sciences Turkey, Gulhane Research and Training Hospital
Locations (1):
- University of Health Sciences Turkey, Gulhane Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kwaan HC. Coronavirus Disease 2019: The Role of the Fibrinolytic System from Transmission to Organ Injury and Sequelae. Semin Thromb Hemost. 2020 Oct;46(7):841-844. doi: 10.1055/s-0040-1709996. Epub 2020 May 9. No abstract available. PMID 32386428